CLINICAL TRIAL: NCT02071732
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Effect on Tinnitus
Brief Title: Therapeutic Effect of Repetitive Transcranial Magnetic Stimulaton on Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Suk Yun Kang, Medical professor, Dongtan Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-002
Record Dates: First submitted 2014-02-19; First posted 2014-02-26 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Patients With Subjective Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real rTMS (Active Comparator): Real rTMS is real continuous theta burst stimulation.
  Interventions: Device: real repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS is sham continuous theta burst stimulation.
  Interventions: Device: sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: real repetitive Transcranial Magnetic Stimulation
  Arms: Real rTMS
Device: sham repetitive Transcranial Magnetic Stimulation — This sham stimulation is not true stimulation.
  Arms: Sham rTMS

SUMMARY:
The purpose of this study is to determine whether repetitive transcranial magnetic stimulation (rTMS) is effective in the treatment of tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjective tinnitus
* Age 18 years and older

Exclusion Criteria:

* Meniere, conductive hearing loss, objective tinnitus
* History of seizure disorder or epilepsy
* Clinically relevant psychiatric comorbidity
* Previous symptomatic stroke
* Surgically or traumatically implanted foreign bodies such as a pacemaker, an implanted medication pump, a metal plate in the skull, or metal inside the skull or eyes (other than dental appliances or fillings), intracardiac lines that may pose a physical hazard during magnetic stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Tinnitus handicap inventory score | Before (- six months) and after (+ 5 days) rTMS interventions
  Primary outcomes will be measured twice. One is before, and the other is after 5-day rTMS interventions. Baseline primary outcome will be acceptable if it is done within the prior 6 months of 1st rTMS. Follow-up primary outcome will be done within the five days after 5th rTMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, and Department of Otorhinolaryngology-Head & Neck Surgery Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea